CLINICAL TRIAL: NCT04362527
Title: Milrinone Infusion for VAsospam Treatment in Subarachnoid hemoRrhage
Acronym: MIVAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019-002145-37
Record Dates: First submitted 2020-04-09; First posted 2020-04-27 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Vasospasm
Keywords: Milrinone
MeSH Terms: interventions — Milrinone; Solutions; Injections; Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Phase 3, multicenter, international (France, Switzerland), randomized, double blinded, placebo-controlled study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Milrinone (Experimental): The patients randomized to this arm will have Milrinone (Laboratoires STRAGEN, France)
  Interventions: Drug: Milrinone 1 Mg/mL Solution for Injection
- Placebo (Placebo Comparator): The patients randomized to this arm will have Saline solution
  Interventions: Drug: Saline solution for injection

INTERVENTIONS:
Drug: Milrinone 1 Mg/mL Solution for Injection — Blinding procedure will be set up for the administration of the treatment
  Other Names: Corotrope
  Arms: Milrinone
Drug: Saline solution for injection — Blinding procedure will be set up for the administration of the treatment
  Other Names: Sodium Chloride 0.9%
  Arms: Placebo

SUMMARY:
Subarachnoid hemorrhage (SAH) is a frequent and severe disease. Mortality can reach 40%. The most frequent complication of SAH is arterial vasospasm, with estimated incidence as high as 70%. Vasospasm is responsible for cerebral ischemia leading to severe morbidity, poorer quality of life and increased mortality.

Intravenous Milrinone, because of vasodilatory properties could be a therapeutic option. We hypothesize that intravenous infusion of Milrinone will improve the neurological recovery of patients with vasospasm following aneurysmal SAH at 3 months.

This is a Phase III, multi-center, randomized, double-blinded, placebo-controlled study. The primary outcome will be the proportion of patients with a good outcome 3 months (defined as a modified rankin score ≤2).

DETAILED DESCRIPTION:
Subarachnoid hemorrhage (SAH) is relatively frequent, accounting for 5% of strokes, and affects a relatively young population. It is essentially caused by cerebral aneurysm rupture. Mortality can reach 40%. The most frequent complication of SAH is arterial vasospasm, with estimated incidence as high as 70%. Vasospasm is responsible for cerebral ischemia, delayed or not, which in turn is responsible for severe morbidity (neurological deficit, neuro psychiatric disorders...), poorer quality of life (institutionalization, inability to return to work ...) and increased mortality.

The pathophysiology of vasospasm is complex, multifactorial and far from being fully understood. Many drugs have been studied in the treatment of symptomatic vasospasm but none has really proven its efficacy. Milrinone is proposed for the treatment of cerebral vasospasm, either as intra-arterial injection (during angiography) or intravenously using continuous infusion. Indeed, among new vasospasm's treatments, Milrinone seems to have good angiographic and clinical results. There is no randomized controlled trials evaluating Milrinone for preventive and/or curative treatment of cerebral vasospasm following aneurysmal SAH. The literature is made only of clinical cases, cases series with angiographic studies or interventional studies not controlled and with no more than 10 patients.

Thus we hypothesize that the intravenous infusion of Milrinone will improve the neurological recovery of patients with vasospasm following aneurysmal SAH at 3 months.

Adult patients, hospitalized for a vasospasm complicating subarachnoid hemorrhage secondary to intracranial aneurysm rupture will be included and randomized within 6 hours of the CT-scanner confirming the vasospasm diagnosis to receive either the study drug (milrinione, a 0,1 mg/kg bolus followed by a 1 μg/kg/min perfusion) or placebo (saline, with a bolus and a continuous infusion). Study drug administration will be formalized (minimum duration 48 hours, maximum duration 14 days).The primary endpoint will be the proportion of patients with a good outcome 3 months (defined as a modified rankin score ≤2).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients hospitalized for aneurysmal SAH
* First episode of vasospasm, with a diagnosis confirmed on cerebral arterial CT-scanner
* Delay between diagnosis of vasospasm (done by CT-scanner) and inclusion ≤6 hours
* Informed consent from a legal representative, or emergency procedure

Exclusion Criteria:

* Initial Glasgow score at 3 with a bilateral mydriasis
* Moribund patient
* Contraindication to Milrinone (notably obstructive cardiomyopathy…)
* Cerebral infarction in the vasospasm area already present on the CT-scanner at the time of diagnosis (lack of expected benefit of treatment in this case according to medical judgement)
* Cardiac failure requiring inotrope administration at the time of randomisation
* Uncontrolled elevated intra-cranial pressure (i.e. ICP>25 mmHg for more than 20 minutes)
* Patient with flutter or cardiac arrhythmia (atrial fibrillation) poorly tolerated
* Major metabolic disturbance (uncorrected hypokalaemia <3 mmol/L)
* Non-affiliation to French health care coverage,
* Pregnant, breastfeeding or parturient woman
* Adult deprived of their liberty by judicial or administrative decision
* Adult under compulsory psychiatric care
* Adult patient protected under the law (guardianship or trusteeship)
* Inclusion in an interventional study using Milrinone, or evaluating a treatment of cerebral vasospasm or with the same primary endpoint (mRS at 3 months).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2025-10-11 (Actual); Study Completion 2026-01-12 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with a good outcome at 3 months | 3 months
  modified Rankin score ≤2 (0 = No symptoms, 1 = No significant disability. Able to carry out all usual activities, despite some symptoms, 2 = Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities, 3 = Moderate disability. Requires some help, but able to walk unassisted, 4 = Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted, 5 = Severe disability. Requires constant nursing care and attention, bedridden, incontinent, 6 = Death)

SECONDARY OUTCOMES:
Mortality rates in intensive care and in hospital | up to 6 months
  To assess mortality rates in intensive care unit and in hospital and 6 months after aneurysm rupture.
Modified Rankin Score at 3 and 6 months | 3 and 6 months
  0 = No symptoms, 1 = No significant disability. Able to carry out all usual activities, despite some symptoms, 2 = Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities, 3 = Moderate disability. Requires some help, but able to walk unassisted, 4 = Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted, 5 = Severe disability. Requires constant nursing care and attention, bedridden, incontinent, 6 = Death
Glasgow outcome scale Extended at 3 and 6 months | up to 6 months
  1= Death, 2=Persistent vegetative state, 3=Sever disability, 4=Moderate disability, 5=Good recovery 2. Persistent vegetative state
  3. Severe disability 4. Moderate disability 5. Low disability
EQ-5D | up to 6 months
  Obtained by centralized telephone interview
Evaluation of the radiologic effectiveness of the treatment | up to 14 days
  Evaluation of the angiographic success according to angiographic CT-scannerwith blind analysis (coted as follows: light success, moderate success or important success)
Evaluation of the radiologic effectiveness of the treatment | 3 months
  Volume of infarcted areas at MRI control if available
Evaluation of the hemodynamic tolerance of the treatment | 24 hours
  need to introduce and/or increase doses of catecholamines by + 50% during the first 24 hours
Evaluation of the metabolic tolerance of the treatment | up to 14 days
  The occurrence of dysnatremia (<135 mmol / L or> 155 mmol / L), Daily diuresis.
cerebral artery flow velocities | H0, H+2, H24+/-12h, H48+/-12h
  Describe treatment-related variations in middle cerebral artery flow velocities.
Length of stay in the intensive care unit and in the hospital | 3 months
  Number of days alive in the intensive care unit and in the hospital
live patient rate | 3 months and 6 months
Describe the number of therapeutic arteriographies | Day 14
  number of artheriographies

CONTACTS AND LOCATIONS:
Overall Officials: Karim KL LAKHAL, PH, Principal Investigator — University Hospital of Nantes; Olivier OH HUET, PU-PH, Principal Investigator — Cavale Blanche - University Hospital of Brest; Pierre-François PP PERRIGAULT, PU-PH, Principal Investigator — Hôpital Gui de Chauliac - University Hospital of Montpellier; Julien JP POTTECHER, PU-PH, Principal Investigator — Hôpital de Hautepierre, University Hospital of Strasbourg; Russel RC CHABANNE, PH, Principal Investigator — Hôpital Gabriel Montpied, University Hospital of Clermont-Ferrand; Benjamin BC Chousterman, PH, Principal Investigator — Hôpital Lariboisière, Paris (AP-HP); Marc ML Laffon, PU-PH, Principal Investigator — Hôpital Bretonneau - University Hospital of Tours; Yoann YL Launey, PH, Principal Investigator — University Hospital of Rennes; Claire CD Dahyot Fizelier, PU-PH, Principal Investigator — University Hospital of Poitiers; Belaid BB Bouhemad, PU-PH, Principal Investigator — University Hospital of Dijon
Locations (16):
- France (16):
  - CHU Angers, Angers
  - CHU Besançon, Besançon
  - CHU Bordeaux, Bordeaux
  - CHU Brest, Brest
  - CHU Caen, Caen
  - Hôpital Gabriel Montpied, Clermont-Ferrand
  - CHU Dijon, Dijon
  - CHU Lille, Lille
  - Hôpital Civils de Lyon, Lyon
  - Hôpital Gui de Chauliac, Montpellier
  - CHU Nantes, Nantes
  - APHP Lariboisière, Paris
  - Hôpital Fondation ROTHSCHILD, Paris
  - CHU Rennes, Rennes
  - Hôpital de Hautepierre, Strasbourg
  - CHU Tours, Tours

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonable request. Only de-identified data will be shared. Any data collected during the study may be shared. The protocol will be shared initially. Other documents may be shared later upon request (e.g., the CRF to allow a collaborator to select the data to which they wish to have access). The recipients of the data will be researchers. The data will be available for any purpose deemed relevant by the MIVAR investigator, based on a protocol provided by the applicant, after verification of obtaining regulatory authorizations, including the favorable opinion of an ethics committee.
Supporting Information: Study Protocol, SAP
Time Frame: The data will be shared after signing a negotiated data transfer contract (data access agreement), for the duration indicated in the contract.
Access Criteria: The data will be made available via secure transfer (sharing platform validated by Angers CHU: BlueFiles or Oodrive).

REFERENCES:
- [Derived] Lasocki S, Lakhal K, de Courson H, Geslain M, Launey Y, Pottecher J, Trouiller P, Laffon M, Gakuba C, Parot-Schinkel E, Hamel JF, Campfort M, Gaillard T; MiVAR study group; ATLANREA group; SFAR research network. Milrinone infusion for vasospasm treatment in subarachnoid haemorrhage: protocol for a double-blind randomised clinical trial - the MiVAR study. BMJ Open. 2025 Oct 28;15(10):e101483. doi: 10.1136/bmjopen-2025-101483. PMID 41151960
- [Derived] Lasocki S, Bruckert V, Campfort M, Leger M, Rineau E. Restrictive transfusion targets the heart now! Insight from the REALITY study. Anaesth Crit Care Pain Med. 2021 Apr;40(2):100854. doi: 10.1016/j.accpm.2021.100854. Epub 2021 Mar 27. No abstract available. PMID 33781988
- See also: Related Info — https://doi.org/10.1136/bmjopen-2025-101483

DOCUMENTS (1):
  • Statistical Analysis Plan: Statistical Analysis Plan (2026-01-15): https://cdn.clinicaltrials.gov/large-docs/27/NCT04362527/SAP_000.pdf